CLINICAL TRIAL: NCT01781455
Title: A Phase I Clinical Study of BBI503 in Adult Patients With Advanced Solid Tumors
Brief Title: A Study of BBI503 in Adult Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBI503-101
Record Dates: First submitted 2013-01-24; First posted 2013-02-01 (Estimated); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Cancer, Advanced Solid Tumors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BBI503 (Experimental)
  Interventions: Drug: BBI503

INTERVENTIONS:
Drug: BBI503

SUMMARY:
This is an open label, single arm dose escalation study of BBI503 in adult patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent must be obtained and documented according to International Conference on Harmonization (ICH)- Good Clinical Practice (GCP), the local regulatory requirements, and permission to use private health information in accordance with the Health Insurance Portability and Accountability Act (HIPPA) prior to study-specific screening procedures
2. A histologically or cytologically confirmed solid tumor that is metastatic, unresectable, or recurrent and for which standard curative or palliative therapies do not exist or are no longer effective.
3. ≥ 18 years of age
4. Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST)
5. Karnofsky performance status ≥ 70%
6. Male or female patients of child-producing potential must agree to use contraception or avoidance of pregnancy measures during the study and for 30 days after the last BBI503 dose
7. Females of childbearing potential must have a negative serum pregnancy test
8. Aspartate transaminase (AST) and alanine transaminase (ALT) < or equal to 1.5 × upper limit of normal (ULN)
9. Hemoglobin (Hgb) ≥ 10 g/dl
10. Total bilirubin < or equal to 1.5 × ULN
11. Creatinine < or equal to 1.5 x ULN or creatinine clearance > 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
12. Absolute neutrophil count < or equal to 1.5 x 10^9/L
13. Platelets ≥ 100 x 10^9/L
14. Life expectancy ≥ 3 months

Exclusion Criteria:

1. Anti-cancer chemotherapy, radiotherapy, immunotherapy, or investigational agents within four weeks of first dose with the exception for a single dose radiation up to 8 Gray (equal to 800 RAD) with palliative intent for pain control up to 14 days before beginning the administration of BBI503
2. Surgery within 4 weeks prior to first dose
3. Any known untreated brain metastases. Treated subjects must be stable for 4 weeks after completion of that treatment, with image documentation required. Patients must have no clinical symptoms from brain metastases and must be either off steroids or on a stable dose of steroids for at least 2 weeks prior to protocol enrollment. Patients with known leptomeningeal metastases are excluded, even if treated.
4. Pregnant or breastfeeding
5. Significant gastrointestinal disorder(s), in the opinion of the Principal Investigator, (e.g., Crohn's disease, ulcerative colitis, extensive gastric resection and small intestinal resection)
6. Unable or unwilling to swallow BBI503 capsules daily
7. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, clinically significant non-healing or healing wounds, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, significant pulmonary disease (shortness of breath at rest or mild exertion), uncontrolled infection or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2012-02; Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events as a Measure of Safety and Tolerability | Adverse events will be assessed at baseline, while the participant is taking BBI503, and for 30 days after stopping therapy. The average length of this duration is expected to be approximately 4 months.
  Assessment of safety of BBI503 by reporting of adverse events and serious adverse events.
Determination of the recommended Phase 2 dose | Up to treatment discontinuation + 30 days with an estimated treatment duration of 4 weeks

SECONDARY OUTCOMES:
Pharmacokinetic profile (Area under the curve) of BBI503 | During the first 28 days of treatment
  Blood sampling to assess the pharmacokinetic profile (Area under the curve) of BBI503.
Pharmacodynamic activity | During the first 28 days of treatment
  Tumor Biopsy(s) to provide information on analysis of the targets and downstream genes/ effect of BBI503 on cancer stem cells through immunohistochemistry.
Anti-tumor activity | Participants will be assessed every eight weeks for anti-tumor activity.
  To assess the preliminary anti-tumor activity of BBI503.

OTHER OUTCOMES:
Progression Free Survival | The time the participant stays on study until progression will be measured and recorded. This is estimated to be approximately 4 months.
Overall Survival | Participant follow-up for overall survival will occur approximately quarterly for the first year the participant is off study, twice during the second year, and once per year thereafter for up to approximately 100 months.
  The time of overall survival will be measured and recorded for each participant.

CONTACTS AND LOCATIONS:
Locations (19):
- United States (18):
  - Mayo Clinic Cancer Center, Scottsdale, Scottsdale, Arizona
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Indiana University, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic Cancer Center, Rochester, Rochester, Minnesota
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Institute for Translational Oncology Research, Greenville Hospital System, Greenville, South Carolina
  - Texas Oncology- Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology- Fort Worth, Fort Worth, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - Cancer Care Centers of South Texas - HOAST, San Antonio, Texas
  - Texas Oncology- Tyler, Tyler, Texas
  - Virginia Cancer Specialists, P.C., Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Yakima Memorial Hostpial/North Star Lodge, Yakima, Washington
- Ottawa Hospital Cancer Centre, Ottawa, Ontario, Canada